CLINICAL TRIAL: NCT02622568
Title: Investigating Veregen ™ 15% Ointment Treatment For Non-facial Verrucae in Pediatric Patients: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Nnenna Agim, Investigating Veregen ™ 15% Ointment Treatment For Non-facial Verrucae in Pediatric Patients: A Pilot Study, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 092014-012
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Verruca, Warts
MeSH Terms: conditions — Warts | interventions — Cryotherapy; green tea extract polyphenone E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryotherapy and Veregen (Active Comparator): Cryotherapy will be performed on the day of first clinic visit according to current standard of care in Children's Medical Center pediatric outpatient dermatology clinic, which consists of two freeze/thaw cycles for maximum of 10 seconds each. Sinecathecins 15% ointment will be prescribed and initiated immediately following the day of first clinic visit. Sinecathecins 15% ointment will be applied to verrucous lesions twice daily. Follow-up clinical visits will be required at 0 weeks, 6 weeks, and 12 weeks. Clinical photos will be taken at each visit. Verrucae will be measured at each visit using a standard ruler. Outcome measures will be numerical reduction in diameter of verruca.
  Interventions: Procedure: Cryotherapy and Veregen
- Veregen only (Experimental): Veregen ™or sinecathecins 15% ointment will be prescribed and initiated immediately following the day of first clinic visit. Veregen ™ or sinecathecins 15% ointment will be applied to verrucous lesions twice daily per current Children's Medical Center protocol. Follow-up clinical visits will be required at 0 weeks, 6 weeks, and 12 weeks. Clinical photos will be taken at each visit. Verrucae will be measured at each visit using a standard ruler. Outcome measures will be numerical reduction in diameter of verruca.
  Interventions: Drug: Veregen only

INTERVENTIONS:
Drug: Veregen only — Topical application of Veregen 15% ointment on affected areas twice daily
  Arms: Veregen only
Procedure: Cryotherapy and Veregen — Cryotherapy followed by topical application of Veregen 15% ointment on affected areas twice daily
  Arms: Cryotherapy and Veregen

SUMMARY:
The purpose of this study is to investigate topical treatment with Veregen™ 15% ointment as a single therapeutic agent and compare it to combination therapy with Veregen ™ 15% ointment and a single destructive treatment by cryotherapy for non-facial verruca vulgaris in the pediatric population. This novel treatment modality may be useful in the pediatric dermatology community offering a less invasive, painless option for treatment of non-facial verruca vulgaris.

DETAILED DESCRIPTION:
The purpose of this study is to investigate topical treatment with Veregen™ 15% ointment as a single therapeutic agent and compare it to combination therapy with Veregen ™ 15% ointment and a single destructive treatment by cryotherapy for non-facial verruca vulgaris in the pediatric population. The investigators will compare the single and combination treatment modalities over identical time points in patients with non-facial verruca vulgaris. One of the current options for care for non-facial verruca includes cryotherapy, which is a painful and destructive method performed in the pediatric dermatology clinic. This study aims to establish the safety, non-invasivenature, efficiency, and efficacy of Veregen ™ 15% ointment as monotherapyfor non-facial verruca vulgaris in the pediatric population. The investigators hypothesize that Veregen ™ 15% ointment monotherapy will non-invasively treat non-facial verruca vulgaris with similar efficacy as combination therapy with a single cryotherapy treatment followed by topical application of Veregen ™ ointment. This novel treatment modality will be useful in the pediatric dermatology community offering a less invasive, painless option for treatment of non-facial verruca vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any ethnic background
* Age between 6 years old and 16 years old
* A clinical diagnosis of non-facial verruca vulgaris
* Able to adhere to study visit schedule, Veregen ™ treatment requirements, and baseline cryotherapy treatment in half of patients
* Verruca size greater than 5 mm

Exclusion Criteria:

* Medically unstable patients
* Patients with immunosuppression
* Families who decline participation
* Verruca may not have been treated in preceding 4 weeks prior to enrollment
* Verruca may not be located on the face or genitalia
* Verruca size less than 5 mm

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UTSW Department of Dermatology, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric Dermatology Medical Clinic
Groups:
- Cryotherapy + Veregen: Cryotherapy will be performed on the day of first clinic visit according to current standard of care in Children's Medical Center pediatric outpatient dermatology clinic, which consists of two freeze/thaw cycles for maximum of 10 seconds each. Veregen ™ 15% ointment will be prescribed and initiated immediately following the day of first clinic visit. Veregen ™ 15% ointment will be applied to verrucous lesions twice daily per current Children's Medical Center protocol. Follow-up clinical visits will be required at 0 weeks, 6 weeks, and 12 weeks. The first day of treatment will begin on the day of first clinic visit (0 weeks). Clinical photos will be taken at each visit. Verrucae will be measured at each visit using a standard ruler. Outcome measures will be numerical reduction in diameter of verruca.
  Veregen or Sinecatechins
- Veregen Only: Veregen ™ 15% ointment will be prescribed and initiated immediately following the day of first clinic visit. Veregen ™ 15% ointment will be applied to verrucous lesions twice daily per current Children's Medical Center protocol. Follow-up clinical visits will be required at 0 weeks, 6 weeks, and 12 weeks. The first day of treatment will begin on the day of first clinic visit (0 weeks). Clinical photos will be taken at each visit. Verrucae will be measured at each visit using a standard ruler. Outcome measures will be numerical reduction in diameter of verruca.
  Veregen or Sinecatechins
Period: Overall Study
Arm/Group | Cryotherapy + Veregen | Veregen Only
Started | 14 | 14
Completed | 9 | 9
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Cryotherapy + Veregen: Cryotherapy will be performed on the day of first clinic visit according to current standard of care in Children's Medical Center pediatric outpatient dermatology clinic, which consists of two freeze/thaw cycles for maximum of 10 seconds each. Veregen ™ 15% ointment will be prescribed and initiated immediately following the day of first clinic visit. Veregen ™ 15% ointment will be applied to verrucous lesions twice daily per current Children's Medical Center protocol. Follow-up clinical visits will be required at 0 weeks, 6 weeks, and 12 weeks. The first day of treatment will begin on the day of first clinic visit (0 weeks). Clinical photos will be taken at each visit. Verrucae will be measured at each visit using a standard ruler. Outcome measures will be numerical reduction in diameter of verruca.
  Veregen or Sinecatechins + cryotherapy
- Total: Total of all reporting groups
Arm/Group | Cryotherapy + Veregen | Veregen Only | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 28
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (3.14) | 10.1 (2.47) | 9.6 (2.79)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Analysis limited to participants that completed the study
  Participants
    number analyzed (Participants) | 9 | 9 | 18
    Female | 3 | 5 | 8
    Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28
Diameter of verrucae at presentation [Mean (Standard Deviation); unit: mm] — Population: Only participants completing study are included in analysis.
  mm
    number analyzed (Participants) | 9 | 9 | 18
    (all) | 6.444 (1.9437) | 6.222 (1.922) | 6.3 (1.88)

OUTCOME MEASURES:

1. Primary Outcome: Size of Verrucae (Warts)
Description: Diameter of verrucae (warts) at week 12
Time Frame: 12 weeks
Population: Only participants completing study are included in analysis.
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Cryotherapy + Veregen: Cryotherapy will be performed on the day of first clinic visit according to current standard of care in Children's Medical Center pediatric outpatient dermatology clinic, which consists of two freeze/thaw cycles for maximum of 10 seconds each. Veregen ™ 15% ointment will be prescribed and initiated immediately following the day of first clinic visit. Veregen ™ 15% ointment will be applied to verrucous lesions twice daily per current Children's Medical Center protocol. Follow-up clinical visits will be required at 0 weeks, 6 weeks, and 12 weeks. The first day of treatment will begin on the day of first clinic visit (0 weeks). Clinical photos will be taken at each visit. Verrucae will be measured at each visit using a standard ruler. Outcome measures will be numerical reduction in diameter of verruca.
  Veregen or Sinecatechins following cryotherapy
Arm/Group | Cryotherapy + Veregen | Veregen Only
Number analyzed (Participants) | 9 | 9
millimeters | 2.333 (3.3541) | 3.889 (3.9826)
Statistical Analysis 1: Comparison: Cryotherapy + Veregen vs Veregen Only; Test type: Non-Inferiority — Veregen alone has efficacy compared to Veregen + cryotherapy; p = 0.383, t-test, 2 sided — Comparison at week 12; Mean Difference (Final Values) = 1.556
Statistical Analysis 2: Comparison: Cryotherapy + Veregen vs Veregen Only; Test type: Non-Inferiority — Comparison at week 0; p = 0.81, t-test, 2 sided; Mean Difference (Final Values) = -0.222

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Cryotherapy + Veregen | Veregen Only
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryotherapy + Veregen (N=14) | Veregen Only (N=14)
Minor irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — transient itching and redness

LIMITATIONS AND CAVEATS:
Attrition rate acceptable for pilot study. Some participants were lost at the first measurement follow-up, others at the second (6 and 12 weeks respectively).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No